CLINICAL TRIAL: NCT02424097
Title: MI Varnish and MI Paste Plus in a Caries Prevention and Remineralization Study
Acronym: GC-WS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GCAmerica-WS
Record Dates: First submitted 2015-04-15; First posted 2015-04-22 (Estimated); Results first posted 2018-12-24 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Dental White Spots; Dental Caries
Keywords: Prevention
MeSH Terms: conditions — Dental Caries | interventions — casein phosphopeptide-amorphous calcium phosphate nanocomplex

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- MI Paste & MI Varnish (Experimental): MI past will be applied by the patient every night; MI varnish will be applied every three months in the office
  Interventions: Drug: CPP-ACP 5% sodium fluoride varnish & 900ppm fluoride paste
- Standard of Care (Active Comparator): Subjects will use at home regal toothpaste every night and F-mouth rinse as recommended
  Interventions: Drug: 1,100pm F-toothpaste and 0.5%NaF rinse

INTERVENTIONS:
Drug: CPP-ACP 5% sodium fluoride varnish & 900ppm fluoride paste — MI Paste & MI Varnish- in-office:
  varnish application once every 3 months; at baseline, at the end of month 3, 6, and 9 (4 applications)
  - at-home: brushing with regular 1,100ppm F-toothpaste, 2x per day and MI Paste Plus, home application after brushing in the evening; 3-5 minutes with in-home application tray
  Arms: MI Paste & MI Varnish
Drug: 1,100pm F-toothpaste and 0.5%NaF rinse — Standard of care at-home:
  Crest tooth brushing 2x per day - (recommendation OTC Fluoride-rinse in the evening at home 1x per day)
  Arms: Standard of Care

SUMMARY:
The objective of this clinical study is to evaluate the efficacy of multiple applications of MI Varnish in combination with MI Paste Plus in caries protection and remineralization in comparison to the use of a control (Crest 1,100ppm Fluoride tooth paste, Fluoride rinse recommendation) in orthodontic patients in a randomized, single blind, prospective, controlled clinical trial over 12 months.

The effect will be measured by white spot lesion regression and prevention as lesion count. Lesions will be scored using the Enamel Decalcification Index (EDI) area evaluation scheme (primary outcome), International Caries Detection and Assessment System (ICDAS), the caries lesion activity criteria (Nyvad criteria; Bente Nyvad, Scandinavian Researcher), and Quantitative Light Fluorescence (QLF, Inspektor Pro, Netherlands)/SOPROLIFE (SOPROLIFE fluorescence camera system, Acteon, France) evaluation in maxillary and mandibular anterior teeth with orthodontic brackets in treatment and control groups.

DETAILED DESCRIPTION:
The study is designed as randomized, single blind, prospective, clinical trial over 12 months. The subjects for this study will be recruited from the University of California at San Francisco UCSF, School of Dentistry, Orthodontic Clinic.

Participants in the study will be patients, who are in orthodontic treatment or will start orthodontic treatment; subjects must have full fixed appliances, with brackets bonded to the buccal surfaces of the maxillary and mandibular incisors, canines and first bicuspids. Subjects will be of moderate or high caries risk according to Caries Risk Assessment and ATP (Adenosine triphosphate) bacteria testing. Subjects will present with at least two active white spot lesions on his/her anterior teeth at the start of the study. The age limitation is ≥ 11 years.

The subjects will be randomly assigned to 1) Experimental group: MI Varnish and MI Paste Plus or 2) Control standard of care group: 1,100 ppm Fluoride tooth paste and recommendation to use OTC (Over-the-counter) Fluoride-rinse in the evening at home.

The clinical study investigator will evaluate the labial/buccal surfaces of upper and lower anterior teeth (first bicuspid to first bicuspid) for white spot lesions (WSL) at baseline and at the end of 3, 6, and 12 months. Newly formed lesions and changes in existing white spot lesions will be documented (using Enamel Decalcification Index (EDI), ICDAS II, light digital photographs and blue fluorescence photography SOPROLIFE and QLF- Quantitative Light Fluorescence).

All subjects will receive one professional tooth cleaning at baseline and at each other evaluation office visit to allow WSL evaluation (cleaning with ultrasonic device, and prophylaxis brush) and treatment application.

ELIGIBILITY:
Inclusion Criteria:

* age 11 or older,
* good health,
* either gender
* present with at least two active white spot lesions on his/her anterior teeth at the start of the study
* have a moderate or high caries risk according to CAMBRA (Caries Management By Risk Assessment) rules
* require at least 12 additional months of full fixed appliance therapy from the time they are recruited for the study
* able to cooperate for treatment in the dental chair and follow at-home instructions
* have an understanding of the study
* willing to comply with all study procedures and protocols
* patient participant is able to provide written informed consent in English; if the participant is a minor, the parent/guardian is able to provide written informed consent in English and the patient participant is able to provide written assent in English
* patient participant or if a minor, the parent/guardian, is willing to sign the "Authorization for Release of Personal Health Information and Use of Personally Unidentified Study Data for Research" form; data will only be used for research
* verifiable records of bonding with Transbond Plus Self-Etching Primer (3M Unitek, Monrovia, CA) and Transbond Light Cure Adhesive or similar products
* verifiable records that "ProSeal" has not been applied at any time during the orthodontic treatment

Exclusion Criteria:

* untreated cavitated lesions
* extensive composite fillings on buccal surfaces of front teeth/first bicuspids or more than one dental crown on front teeth/first bicuspids
* has sealants or fluoride releasing cements on the buccal surface of the anterior teeth
* in-office fluoride treatment in the last three months
* history of using any products containing CCP-ACP (casein phosphopeptides and amorphous calcium phosphate; MI paste, chewing gums or candies, etc.), prescription Fluoride products, and Chlorhexidine use in the last three months
* intrinsic or extremely heavy extrinsic staining
* any signs of fluorosis in the dentition
* any signs of morphologic/anatomical/developmental deviations in the teeth
* previous history of in office bleaching treatment
* subject not willing to stop the use of any other oral hygiene product than those prescribed/suggested
* has underlying systemic disease which could alter enamel composition or formation
* suffering from systemic diseases, significant past or medical history with conditions that may affect oral health or oral flora (i.e. diabetes, HIV, heart conditions that require antibiotic prophylaxis)
* use of medication causing dry mouth (extreme high caries risk)
* subject is pregnant or lactating
* milk protein allergy
* any illness/condition that the investigator feels will affect the study outcome
* will leave the area and will not be available for recall visits
* subjects who are not willing to inform us about prospective visits of other dentist and will not allow us to discuss treatment with those dentist
* subjects who are not willing to refrain from any additional professional tooth cleaning or any additional Fluoride application.

Min Age: 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-05; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Rechmann, DMD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF School of Dentistry - Dental Offices in Bay Area, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mitchell L. Decalcification during orthodontic treatment with fixed appliances--an overview. Br J Orthod. 1992 Aug;19(3):199-205. doi: 10.1179/bjo.19.3.199. No abstract available. PMID 1390575
- [Result] Geiger AM, Gorelick L, Gwinnett AJ, Griswold PG. The effect of a fluoride program on white spot formation during orthodontic treatment. Am J Orthod Dentofacial Orthop. 1988 Jan;93(1):29-37. doi: 10.1016/0889-5406(88)90190-4. No abstract available. PMID 3276146
- [Result] Richter AE, Arruda AO, Peters MC, Sohn W. Incidence of caries lesions among patients treated with comprehensive orthodontics. Am J Orthod Dentofacial Orthop. 2011 May;139(5):657-64. doi: 10.1016/j.ajodo.2009.06.037. PMID 21536209
- [Result] Magness WS, Shannon IL, West DC. Office-applied fluoride treatments for orthodontic patients. J Dent Res. 1979 Apr;58(4):1427. doi: 10.1177/00220345790580042401. No abstract available. PMID 285114
- [Result] Stratemann MW, Shannon IL. Control of decalcification in orthodontic patients by daily self-administered application of a water-free 0.4 per cent stannous fluoride gel. Am J Orthod. 1974 Sep;66(3):273-9. doi: 10.1016/0002-9416(74)90291-7. No abstract available. PMID 4528489
- [Result] Mizrahi E. Surface distribution of enamel opacities following orthodontic treatment. Am J Orthod. 1983 Oct;84(4):323-31. doi: 10.1016/s0002-9416(83)90348-2. PMID 6605091
- [Result] Gorelick L, Geiger AM, Gwinnett AJ. Incidence of white spot formation after bonding and banding. Am J Orthod. 1982 Feb;81(2):93-8. doi: 10.1016/0002-9416(82)90032-x. PMID 6758594
- [Result] Zachrisson BU, Zachrisson S. Caries incidence and oral hygiene during orthodontic treatment. Scand J Dent Res. 1971;79(6):394-401. doi: 10.1111/j.1600-0722.1971.tb02028.x. No abstract available. PMID 5288673
- [Result] Gorton J, Featherstone JD. In vivo inhibition of demineralization around orthodontic brackets. Am J Orthod Dentofacial Orthop. 2003 Jan;123(1):10-4. doi: 10.1067/mod.2003.47. PMID 12532056
- [Result] Zachrisson BU. Fluoride application procedures in orthodontic practice, current concepts. Angle Orthod. 1975 Jan;45(1):72-81. doi: 10.1043/0003-3219(1975)0452.0.CO;2. PMID 1054935
- [Result] Geiger AM, Gorelick L, Gwinnett AJ, Benson BJ. Reducing white spot lesions in orthodontic populations with fluoride rinsing. Am J Orthod Dentofacial Orthop. 1992 May;101(5):403-7. doi: 10.1016/0889-5406(92)70112-N. PMID 1590288
- [Result] Benson PE, Parkin N, Millett DT, Dyer FE, Vine S, Shah A. Fluorides for the prevention of white spots on teeth during fixed brace treatment. Cochrane Database Syst Rev. 2004;(3):CD003809. doi: 10.1002/14651858.CD003809.pub2. PMID 15266503
- [Result] Ogaard B, Alm AA, Larsson E, Adolfsson U. A prospective, randomized clinical study on the effects of an amine fluoride/stannous fluoride toothpaste/mouthrinse on plaque, gingivitis and initial caries lesion development in orthodontic patients. Eur J Orthod. 2006 Feb;28(1):8-12. doi: 10.1093/ejo/cji075. Epub 2005 Oct 17. PMID 16230329
- [Result] Andersson A, Skold-Larsson K, Hallgren A, Petersson LG, Twetman S. Effect of a dental cream containing amorphous cream phosphate complexes on white spot lesion regression assessed by laser fluorescence. Oral Health Prev Dent. 2007;5(3):229-33. PMID 17977295
- [Result] Beerens MW, van der Veen MH, van Beek H, ten Cate JM. Effects of casein phosphopeptide amorphous calcium fluoride phosphate paste on white spot lesions and dental plaque after orthodontic treatment: a 3-month follow-up. Eur J Oral Sci. 2010 Dec;118(6):610-7. doi: 10.1111/j.1600-0722.2010.00780.x. PMID 21083623
- [Result] Reynolds EC. Remineralization of enamel subsurface lesions by casein phosphopeptide-stabilized calcium phosphate solutions. J Dent Res. 1997 Sep;76(9):1587-95. doi: 10.1177/00220345970760091101. PMID 9294493
- [Result] Oshiro M, Yamaguchi K, Takamizawa T, Inage H, Watanabe T, Irokawa A, Ando S, Miyazaki M. Effect of CPP-ACP paste on tooth mineralization: an FE-SEM study. J Oral Sci. 2007 Jun;49(2):115-20. doi: 10.2334/josnusd.49.115. PMID 17634723
- [Result] Sudjalim TR, Woods MG, Manton DJ, Reynolds EC. Prevention of demineralization around orthodontic brackets in vitro. Am J Orthod Dentofacial Orthop. 2007 Jun;131(6):705.e1-9. doi: 10.1016/j.ajodo.2006.09.043. PMID 17561043
- [Result] Cai F, Shen P, Morgan MV, Reynolds EC. Remineralization of enamel subsurface lesions in situ by sugar-free lozenges containing casein phosphopeptide-amorphous calcium phosphate. Aust Dent J. 2003 Dec;48(4):240-3. doi: 10.1111/j.1834-7819.2003.tb00037.x. PMID 14738126
- [Result] Uysal T, Amasyali M, Ozcan S, Koyuturk AE, Akyol M, Sagdic D. In vivo effects of amorphous calcium phosphate-containing orthodontic composite on enamel demineralization around orthodontic brackets. Aust Dent J. 2010 Sep;55(3):285-91. doi: 10.1111/j.1834-7819.2010.01236.x. PMID 20887516
- [Result] Wang JX, Yan Y, Wang XJ. Clinical evaluation of remineralization potential of casein phosphopeptide amorphous calcium phosphate nanocomplexes for enamel decalcification in orthodontics. Chin Med J (Engl). 2012 Nov;125(22):4018-21. PMID 23158136
- [Result] Robertson MA, Kau CH, English JD, Lee RP, Powers J, Nguyen JT. MI Paste Plus to prevent demineralization in orthodontic patients: a prospective randomized controlled trial. Am J Orthod Dentofacial Orthop. 2011 Nov;140(5):660-8. doi: 10.1016/j.ajodo.2010.10.025. PMID 22051486
- [Result] Huang GJ, Roloff-Chiang B, Mills BE, Shalchi S, Spiekerman C, Korpak AM, Starrett JL, Greenlee GM, Drangsholt RJ, Matunas JC. Effectiveness of MI Paste Plus and PreviDent fluoride varnish for treatment of white spot lesions: a randomized controlled trial. Am J Orthod Dentofacial Orthop. 2013 Jan;143(1):31-41. doi: 10.1016/j.ajodo.2012.09.007. PMID 23273358
- [Result] Bader JD. Casein phosphopeptide-amorphous calcium phosphate shows promise for preventing caries. Evid Based Dent. 2010;11(1):11-2. doi: 10.1038/sj.ebd.6400701. PMID 20348890
- [Result] Nyvad B, Machiulskiene V, Baelum V. Reliability of a new caries diagnostic system differentiating between active and inactive caries lesions. Caries Res. 1999 Jul-Aug;33(4):252-60. doi: 10.1159/000016526. PMID 10343087
- [Result] Terrer E, Koubi S, Dionne A, Weisrock G, Sarraquigne C, Mazuir A, Tassery H. A new concept in restorative dentistry: light-induced fluorescence evaluator for diagnosis and treatment. Part 1: Diagnosis and treatment of initial occlusal caries. J Contemp Dent Pract. 2009 Nov 1;10(6):E086-94. PMID 20020086
- [Result] Rechmann P, Charland D, Rechmann BM, Featherstone JD. Performance of laser fluorescence devices and visual examination for the detection of occlusal caries in permanent molars. J Biomed Opt. 2012 Mar;17(3):036006. doi: 10.1117/1.JBO.17.3.036006. PMID 22502564

RESULTS

PARTICIPANT FLOW:
Groups:
- MI Paste & MI Varnish: MI past will be applied by the patient every night; MI varnish will be applied every three months in the office
  CPP-ACP 5% sodium fluoride varnish & 900ppm fluoride paste: MI Paste & MI Varnish- in-office:
  varnish application once every 3 months; at baseline, at the end of month 3, 6, and 9 (4 applications)
  - at-home: brushing with regular 1,100ppm F-toothpaste, 2x per day and MI Paste Plus, home application after brushing in the evening; 3-5 minutes with in-home application tray
Period: Overall Study
Arm/Group | MI Paste & MI Varnish | Standard of Care
Started | 20 | 20
Completed | 19 | 18
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MI Paste & MI Varnish | Standard of Care | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 17 | 17 | 34
  Between 18 and 65 years | 3 | 3 | 6
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.1 (3.8) | 16.5 (3.8) | 16.1 (3.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 19
  Male | 9 | 12 | 21
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Change in White Spot Lesions Count - Enamel Decalcification Index (EDI)
Description: The area evaluation scheme of the Enamel Decalcification Index (EDI) divides the buccal surface of each tooth into 4 quadrants and then registers the possible existence of a white spot lesion (decalcification) in each of these 4 quadrants. For each quadrant the lesion can be scaled as: 0 = no decalcification, 1 = decalcification covering <50% of the area, 2 = decalcification covering > 50% of the area, 3 = decalcifications covering 100% of the area or severe decalcification with cavitation. Thus, for each tooth the value can range between 0 and 12.
  16 teeth per subject were evaluated, for each subject the value of each tooth was added - thus the range per one subject can be between 0 and 192.
  A mean over all participants in one group was calculated. A higher score means a worse outcome.
Time Frame: Baseline and 12-months
Population: enamel decalcification index (EDI)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MI Paste & MI Varnish | Standard of Care
Number analyzed (Participants) | 19 | 18
units on a scale | 40.2 (13.6) | 41.3 (11.8)

2. Secondary Outcome: Change in International Caries Detection and Assessment System (ICDAS II) to Score for Smooth Surfaces White Spot Lesions (WSL)
Description: The International Caries Detection and Assessment System (ICDAS II) is a standardized method of caries lesion assessment.The score is based on apparent lesion severity, with scores from 0 to 6.The buccal surface of each tooth was divided into 4 quadrants, and for each quadrant a score was assigned with ICDAS scores: 0 = sound, 1 = first visual change in enamel, after air drying, 2 = distinct demineralization visual change in enamel, 3 = localized enamel breakdown due to caries with no visible dentin, 4 = surface with underlying dark shadow from dentin with or without enamel breakdown, 5 = distinct cavity with visible dentin, 6 = extensive cavity with visible dentin.
  The ICDAS scores were calculated as the sum of the highest ICDAS scores assigned to each examined tooth per subject. 16 teeth per subject were evaluated, thus, for each subject the value can range between 0 and 96.
  A mean over all participants in one group was calculated. A higher score means a worse outcome.
Time Frame: Baseline and 12-months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MI Paste & MI Varnish | Standard of Care
Number analyzed (Participants) | 19 | 18
score on a scale | 22.3 (5.9) | 22.6 (4.9)

3. Other Pre Specified Outcome: Change in Lesion Activity, Nyvad Criteria
Description: WS lesion activity will be determined using the Nyvad criteria;
Time Frame: Baseline and 12-months
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Change in SOPROLIFE
Description: fluorescence measurements using blue light fluorescence make WSLs visible for scoring;
Time Frame: Baseline and 12-months
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Change in Quantitative Light Fluorescence (QLF)
Description: Quantitative Light Fluorescence will be used to evaluate the WSL
Time Frame: Baseline and 12-months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year, 8 months
Arm/Group | MI Paste & MI Varnish | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No